CLINICAL TRIAL: NCT00835159
Title: Rivastigmine in the Treatment of Postoperative Delirium: a Pilot Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H# 08-765
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction
Keywords: Postoperative Delirium; Postoperative Cognitive Dysfunction; Rivastigmine; Exelon; Memory impairment; Delirium; Cognitive function
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications; Emergence Delirium; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivastigmine Patch (Experimental): Group receiving Rivastigmine Patch
  Interventions: Drug: Rivastigmine Patch
- Placebo Patch (Placebo Comparator): A 2x2 gauze and a Tegaderm dressing applied to upper back within 3 hours of surgery for a period of 24 hours.
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: Rivastigmine Patch — Rivastigmine Patch 4.6 mg/24 hours: 5 cm2 size containing 9 mg rivastigmine applied to upper back preoperatively for a period of 24 hours
  Other Names: Exelon Patch
  Arms: Rivastigmine Patch
Other: Placebo Patch — A 2x2 gauze and a Tegaderm dressing applied to upper back within 3 hours of surgery for a period of 24 hours.
  Arms: Placebo Patch

SUMMARY:
The purpose of this study is to determine whether preoperative administration of Rivastigmine prevents the incidence of postoperative delirium in patients undergoing major surgery as well as postoperative cognitive dysfunction.

DETAILED DESCRIPTION:
Postoperative delirium (POD) and Postoperative cognitive dysfunction (POCD) are common significant postoperative complications in elderly patients. A reduction of postoperative complications would lead to improved functional status, greater independence and reduction in health care cost. Scientific evidence shows that acetylcholinesterase inhibitors may reduce incidence and/or severity of postoperative delirium. We propose to conduct a randomized, double-masked, placebo-controlled study to assess effectiveness of Rivastigmine, an acetylcholinesterase inhibitor. Rivastigmine transdermal system (Exelon Patch) is approved by FDA for the treatment of mild to moderate Alzheimer's dementia and mild to moderate dementia associated with Parkinson's disease. Patients 65 y.o. and older undergoing major elective surgery will qualify for the study based on risk assessment guidelines. Patients screening will include Mini Mental Status Examination (MMSE to assess baseline cognitive function), Hamilton scale (to screen for depression), Telephone Interview of Cognitive Status Modified (TICS-M to assess baseline cognitive function over the phone) and Brief Test of Adult Cognition by Telephone (BTACT to assess baseline cognitive function over the phone). All study subjects will be randomly assigned to one of 2 groups prior to surgery. The treatment group will receive a Rivastigmine patch preoperatively covered by tegaderm dressing and a placebo group will receive just a tegaderm dressing. Both groups will be assessed twice daily at 9am and 4pm for up to 72 hours postoperatively with Confusion Assessment Method for Intensive Care Unit (CAM-ICU), Memorial Delirium Assessment Scale (MDAS) and Mini Mental Status Examination (to diagnose delirium and assess its severity). At one month and three months postoperatively subjects with a postoperative MMSE of 27 or less will be assessed for postoperative cognitive dysfunction. The assessment will be performed over the phone with TICS-M and Brief Test of Adult Cognition by Telephone. Outcomes will be divided into Primary and Secondary outcomes. Primary outcome will determine the proportions of patients with at least one episode of POD in the treatment and placebo groups, diagnosed by CAM-ICU. Secondary outcome will determine the proportions of patients with development of POCD in both groups, diagnosed by TICS-M at 1 month postoperatively. Secondary outcome will also determine cumulative number of POD episodes within first 3 days of hospital stay as diagnosed by CAM-ICU, severity of POD as diagnosed by the MDAS, recovery of cognitive function as diagnosed by MMSE, TICS-M and BTACT, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

65 ≥ y.o. undergoing major elective surgery over 2 hours in length with one or more of the following:

* Preoperative cognitive impairment
* Age > 70 y.o.
* Use of psychoactive medications
* History of prior delirium
* Severe illness/co-morbidity

Exclusion Criteria:

* Delirium on admission Profound dementia No spoken/written English An emergent procedure Hypersensitivity to Rivastigmine

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bekker, MD, PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, Department of Anesthesiology 550 First Avenue, RR-603, New York, New York, United States

REFERENCES:
- [Result] Zaslavsky A, Haile M, Kline R, Iospa A, Frempong-Boadu A, Bekker A. Rivastigmine in the treatment of postoperative delirium: a pilot clinical trial. Int J Geriatr Psychiatry. 2012 Sep;27(9):986-8. doi: 10.1002/gps.2801. No abstract available. PMID 22886871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patientsof 65years and older admitted for elective surgery undergeneral anesthesia were screened. Only patients at risk fordeveloping POD were considered for recruitment
Pre-assignment Details: This was a randomized, placebo controlled, double-blind clinical trial. Screened patients were 65 years +, having elective surgery under general anesthesia. Only patients at risk for POD were considered for recruitment. Eligible patients received rivastigmine 5cm2 transdermal or placebo patch. 30 patients recruited but only 28 had complete data.
Groups:
- Rivastigmine 5-cm2 Transdermal Patch: Only patients at risk for developing POD were considered for recruitment. That risk was based on the presence of at least one of five predictive factors: (1) preoperative cognitive impairment (Mini mental state examination (MMSE)<24); (2) advanced age (>70 years); (3) preoperative use of psychoactive drugs; (4) history of prior delirium; and/or (5) severe illness or comorbidity. Eligible patients received a rivastigmine 5-cm2 transdermal patch
- Placebo Patch: Only patients at risk for developing POD were considered for recruitment. That risk was based on the presence of at least one of five predictive factors: (1) preoperative cognitive impairment (Mini mental state examination (MMSE)<24); (2) advanced age (>70 years); (3) preoperative use of psychoactive drugs; (4) history of prior delirium; and/or (5) severe illness or comorbidity. Eligible patients received a placebo patch.
Period: Overall Study
Arm/Group | Rivastigmine 5-cm2 Transdermal Patch | Placebo Patch
Started | 11 | 17
Completed | 11 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine 5-cm2 Transdermal Patch | Placebo Patch | Total
Number analyzed (Participants) | 11 | 17 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 11 | 17 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.0909 (5.55796) | 72.6471 (6.52822) | 72.4286 (6.06403)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 11 | 17 | 28

OUTCOME MEASURES:

1. Primary Outcome: Incidence of POD
Description: Is the incidence of POD not affected by rivastigmine treatment or not.
Time Frame: 72 hours postoperatively
Measure: Number; unit: participants
Groups:
- Rivastigmine Patch: Eligible patients received a rivastigmine 5-cm2 transdermal patch
- Placebo Patch: Eligible patients received a placebo patch
Arm/Group | Rivastigmine Patch | Placebo Patch
Number analyzed (Participants) | 11 | 17
participants | 2 | 4

ADVERSE EVENTS:
Time Frame: No adverse events related to the use of a rivastigmine transdermal patch were determined in this clinical trial.
Arm/Group | Rivastigmine 5-cm2 Transdermal Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/17
Other Adverse Events (participants affected / at risk) | 0/11 | 0/17

LIMITATIONS AND CAVEATS:
The study was halted prematurely because of a warning letter issued by the rivastigmine manufacturer indicating the possibility of increased mortality associated with the oral administration of the drug in critically ill patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No